CLINICAL TRIAL: NCT01653418
Title: A Phase II Study of V-BEAM (Bortezomib, Carmustine, Etoposide, Cytarabine, and Melphalan) as Conditioning Regimen Prior to Second Autologous Stem Cell Transplantation for Multiple Myeloma
Brief Title: Phase II Study of V-BEAM Conditioning Regimen Prior to Second Autologous Stem Cell Transplantation
Acronym: V-BEAM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the high rate of morbidity and mortality
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201208046
Record Dates: First submitted 2012-07-23; First posted 2012-07-31 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Carmustine; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- V-BEAM + Stem Cell Infusion (Experimental): Bortezomib IV or SC (1.3mg/m2) on Days -6, -3, +1 and +4 Carmustine IV (300mg/m2) on Day -7 Etoposide IV twice daily (100 mg/m2) on Days -6, -5, -4, and -3 Cytarabine IV twice daily (100 mg/m2) on Days -6, -5, -4, and -3 Melphalan IV (140 mg/m2) on Day-2 Stem cell infusion on Day 0
  Interventions: Drug: Bortezomib; Drug: Carmustine; Drug: Etoposide; Drug: Cytarabine; Drug: Melphalan; Procedure: Stem cell infusion

INTERVENTIONS:
Drug: Bortezomib
  Other Names: Velcade
Drug: Carmustine
  Other Names: BCNU, BiCNU®
Drug: Etoposide
  Other Names: Vepesid, VP-16
Drug: Cytarabine
  Other Names: Ara-C, Cytosar-U, 1-β-Arabinofuranosylcytosine, Arabinosylcytosine, Cytosine arabinoside
Drug: Melphalan
  Other Names: Alkeran®, L-PAM
Procedure: Stem cell infusion

SUMMARY:
BEAM regimen (BCNU, etoposide, cytarabine, and melphalan) is the most commonly used conditioning regimen for relapsed/refractory lymphoma patients needing autologous stem cell transplantation. Since these components are all effective in myeloma and bortezomib has shown promising results in the transplant setting, here the investigators propose a phase II study to investigate the combination of bortezomib and BEAM as a new conditioning regimen for patients who relapse or progress after the first autologous transplantation and for whom a second autologous transplant is considered.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically confirmed diagnosis of multiple myeloma.
* Patient must have received a prior autologous stem cell transplantation with melphalan conditioning for multiple myeloma with subsequent disease progression and repeat autologous stem cell transplantation is deemed appropriate by the treating physicians.
* Patient must receive induction chemotherapy including 2 to 4 cycles of anti-myeloma therapy including bortezomib, with or without immune modulating agents and/or corticosteroids, Completion of induction therapy will occur within 30 days of first study drug dose.
* Patient must have ≥ 2x106/kg CD34+ autologous stem cells available for transplantation.
* Patient must be ≥ 18 years of age.
* Patient must have life expectancy of greater than 6 months.
* Patient must have an ECOG performance status ≤ 2 or Karnofsky performance status ≥ 60% (see Appendices A and B)
* Patient must have normal bone marrow and organ function as defined below within 14 days prior to first study drug dose (conditioning regimen):

  * Absolute neutrophil count ≥500/mm3
  * Platelets ≥ 50,000/mm3
  * Hemoglobin ≥ 8 g/dl
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine clearance (Appendix C) ≥30 mL/min/1.73m2
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry through Day +100 visit. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patient must be able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Patient must not be refractory to induction therapy. Refractory is defined as disease progression while on therapy or within 30 days following completion of therapy.
* Patient must not have had disease progression requiring active treatment within 12 months of previous autologous stem cell transplant. Maintenance therapy is not considered active treatment.
* Patient must not have peripheral neuropathy ≥ grade 3 based on NCI CTCAE v 4.0 (Appendix D).
* Patient must not be receiving renal replacement therapy, hemodialysis, or peritoneal dialysis.
* Patient must not have another concurrent malignancy requiring treatment.
* Patient must not be receiving any other investigational agents within 14 days prior to the first dose of study drug.
* Patient must not have known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib, carmustine, etoposide, cytarabine, and melphalan, or other agents used in the study.
* Patient must not have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient must not be pregnant and/or breastfeeding.

Inclusion of Women and Minorities

-Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 09/20/2012 and closed to participant enrollment on 06/18/2013.
Period: Overall Study
Arm/Group | V-BEAM + Stem Cell Infusion
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | V-BEAM + Stem Cell Infusion
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 64.5 [48 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10
Durie-Salmon Stage of Myeloma on Diagnosis [Number; unit: participants] — STAGE I
  * Hemoglobin >10g/dL
  * Serum calcium normal or <10.5mg/dL
  * Bone x-ray, normal bone structure (scale 0), or solitary bone plasmacytoma only
  * Low M-component production rates IgG value <5g/dL; IgA value <3g/dL
  * Urine light chain M-component on electrophoresis <4g/24h
  STAGE II -Neither Stage I or Stage III
  STAGE III
  * Hemoglobin <8.5g/dL
  * Serum calcium >12mg/dL
  * Advanced lytic bone lesions (scale 3) -High M-component production rates IgG value >7g/dL IgA value >5g/dL- Bence Jones protein >12g/24h
  SUBCLASS
  -A: relatively normal renal function (serum creatinine) <2.0 mg/dL
  participants
    Stage I | 0
    Stage IIA | 3
    Stage IIIA | 7
International Staging System (ISS) Stage of Myeloma on Diagnosis [Number; unit: participants] — STAGE I
  -Serum beta-2 microglobulin is less than 3.5 (mg/L) and the albumin level is above 3.5 (g/L)
  STAGE II -Neither stage I or III
  STAGE III
  -Serum beta-2 microglobulin is greater than 5.5
  participants
    Stage I | 2
    Stage II | 5
    Stage III | 2
    Unknown | 1
Monoclonal Protein Type [Number; unit: participants] — Antibodies typically consist of 2 heavy chains and 2 light chains. There are 5 kinds of heavy chains termed IgG, IgA, IgM, IgD, and IgE; and 2 distinct types of light chain, termed kappa and lambda. In myeloma, all the abnormal plasma cells make the same antibody. Therefore the myeloma can be classified by the type of light and heavy chains produced, such as IgG kappa, IgG lambda, IgA kappa, or IgA lambda, etc.
  Occasionally, the malignant plasma cells make only the light chain component of the antibody. These patients are said to have "light chain myeloma."
  participants
    IgG | 3
    IgA | 5
    Light chain only | 2
Time to Progression from First Transplant [Median (Full Range); unit: months] | 29 [17 to 97]
Time from Diagnosis to V-BEAM transplant [Median (Full Range); unit: months] | 42 [27 to 118]
Number of Prior Therapies (including prior transplant) [Median (Full Range); unit: prior therapies] | 4 [3 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (Complete Response + Stringent Complete Response)
Description: Defined by the International Myeloma Working Group (IMWG) criteria
Time Frame: Day +100
Population: Two participants without evaluable responses due to early mortality were not included in this analysis.
Measure: Number; unit: participants
Arm/Group | V-BEAM + Stem Cell Infusion
Number analyzed (Participants) | 8
participants | 6

2. Secondary Outcome: Number of Participants With Progression-free Survival (PFS)
Description: PFS is defined as the duration from transplant to time of first progression, death, relapse after CR, or the date the patient was last known to be in remission.
  Response will be assessed per the International Myeloma Working Group (IMWG) Response Criteria.
Time Frame: Median follow-up of 6 months (range: 6.0-12.0 months)
Population: Two participants without evaluable responses due to early mortality were not included in this analysis.
Measure: Number; unit: participants
Arm/Group | V-BEAM + Stem Cell Infusion
Number analyzed (Participants) | 8
participants
  No relapse/progression | 7
  Relapse/progression at 12 months | 1

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR includes Partial Response (PR) + Very Good Partial Response (VGPR) + Complete Response (CR)
  Response will be assessed per the International Myeloma Working Group (IMWG) Response Criteria.
Time Frame: 3 months following Day +100 visit
Population: Two participants without evaluable responses due to early mortality were not included in this analysis.
Measure: Number; unit: participants
Arm/Group | V-BEAM + Stem Cell Infusion
Number analyzed (Participants) | 8
participants
  Partial response | 0
  Very good partial response | 2
  Complete response | 6

4. Secondary Outcome: Very Good Partial Response Rate (VGPR+nCR+sCR+CR)
Description: Response will be assessed per the International Myeloma Working Group (IMWG) Response Criteria.
Time Frame: Day +100
Population: Two participants without evaluable responses due to early mortality were not included in this analysis.
Measure: Number; unit: participants
Arm/Group | V-BEAM + Stem Cell Infusion
Number analyzed (Participants) | 8
participants | 8

5. Secondary Outcome: Toxicity of V-BEAM
Description: Graded per the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  Patients are evaluated from first receiving study treatment until a 30-day follow-up after the conclusion of treatment for adverse events not resulting in death. Adverse events resulting in death will be evaluated through Day +100.
  This outcomes measures the common toxicities observed. Please refer to the Serious Adverse Event and Other Adverse Event sections of the results for further details.
Time Frame: 30 days after end of treatment / Day +100
Measure: Number; unit: participants
Arm/Group | V-BEAM + Stem Cell Infusion
Number analyzed (Participants) | 10
participants
  Neutropenic fever | 10
  Clostridium difficile colitis | 3
  Neutropenic colitis without Clostridium difficile | 3
  Sepsis | 3
  Mucositis (grade 1-2) | 8
  Mucositis (grade 3-4) | 2
  Diarrhea (grade 3-4) | 10
  Hepatic toxicity (grade 3-4) | 1
  Peripheral neuropathy (grade 1-2) | 2
  Toxic death | 2

6. Secondary Outcome: Time to Neutrophil Engraftment After V-BEAM.
Description: Time to neutrophil engraftment is defined as duration between Day 0 to the first day of ANC > 0.5x109/L post transplant when it is sustained for more than three consecutive days.
Time Frame: Day +100
Population: Two participants without evaluable responses due to early mortality were not included in this analysis.
Measure: Median (Full Range); unit: days
Arm/Group | V-BEAM + Stem Cell Infusion
Number analyzed (Participants) | 8
days | 10 [9 to 11]

7. Secondary Outcome: Number of Participants With Overall Survival (OS)
Description: OS is defined as the duration from the time of transplant to death or last follow-up.
Time Frame: Median follow-up of 6 months (range: 6-12 months)
Measure: Number; unit: participants
Arm/Group | V-BEAM + Stem Cell Infusion
Number analyzed (Participants) | 10
participants
  Expired Day +3 | 1
  Expired Day +18 | 1
  Alive | 8

8. Secondary Outcome: Treatment Related Mortality (TRM) of V-BEAM
Time Frame: Day +100
Measure: Number; unit: participants
Arm/Group | V-BEAM + Stem Cell Infusion
Number analyzed (Participants) | 10
participants | 2

9. Secondary Outcome: Time to Platelet Engraftment After V-BEAM.
Description: Time to platelet engraftment is defined as the duration between Day 0 to the first day of platelet count sustained at > 20x109/L without transfusion. The median time to neutrophil and platelet engraftment will be reported.
Time Frame: Day +100
Population: Two participants without evaluable responses due to early mortality were not included in this analysis.
Measure: Median (Full Range); unit: days
Arm/Group | V-BEAM + Stem Cell Infusion
Number analyzed (Participants) | 8
days
  More than 20 x 10^9/L | 22.5 [17 to 36]
  More than 50 x 10^9/L | 23 [17 to 46]

ADVERSE EVENTS:
Time Frame: Patients are evaluated from first receiving study treatment until a 30-day follow-up after the conclusion of treatment for adverse events not resulting in death. Adverse events resulting in death will be evaluated through Day +100.
Arm/Group | V-BEAM + Stem Cell Infusion
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V-BEAM + Stem Cell Infusion (N=10)
Diarrhea (Gastrointestinal disorders) | 1
Febrile neutropenia (Infections and infestations) | 1
Multi-organ failure (General disorders) | 1
Sepsis (death) (Infections and infestations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | V-BEAM + Stem Cell Infusion (N=10)
Acute gout attack (Musculoskeletal and connective tissue disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Alanine aminotransferase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 10
Aspartate aminotransferase increased (Investigations) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Blood bilirubin increased (Investigations) | 2
Cachexia (Metabolism and nutrition disorders) | 1
Clostridium difficile positive colitis (Infections and infestations) | 3
Creatinine increased (Investigations) | 4
Diarrhea (Gastrointestinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Edema - limbs (General disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 3
Esophageal infection (Infections and infestations) | 1
Febrile neutropenia (Infections and infestations) | 9
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Group B strep bacteremia (Infections and infestations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 10
Hypotension (Vascular disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 10
Mucositis - oral (Gastrointestinal disorders) | 10
Neutrophil count decreased (Investigations) | 10
Peripheral sensory neuropathy (Nervous system disorders) | 2
Platelet count decreased (Investigations) | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Rash (maculo-papular) (Skin and subcutaneous tissue disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Typhlitis (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 10

LIMITATIONS AND CAVEATS:
2 early deaths caused a concern for safety and resulted in suspension of enrollment in May 2013. After a review of the data, the investigators determined that this regimen had unexpected toxicity & the trial was closed to enrollment in June 2013.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes